CLINICAL TRIAL: NCT00706966
Title: A Pilot Study of MRI and Spectroscopy Imaging Changes With 6-months of Dutasteride in Patients With Symptomatic Benign Prostatic Hypertrophy and Low-risk Prostate Cancer on Watchful Waiting or Requiring Neoadjuvant Androgen Suppression Prior to Prostate Brachytherapy
Brief Title: MRI and Magnetic Resonance Spectroscopy Imaging in Patients Receiving Dutasteride for Benign Prostatic Hypertrophy and Low-Risk Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000596822; UCSF-05551 (Other: UCSF); H7056-26910-03 (Other: Committee on Human Research (CHR))
Record Dates: First submitted 2008-06-27; First posted 2008-06-30 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Nonmalignant Neoplasm; Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; benign prostatic hyperplasia
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dutasteride (Experimental): Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months
  Interventions: Drug: dutasteride

INTERVENTIONS:
Drug: dutasteride — 6 months of dutasteride 3.5 mg daily
  Other Names: Avodart

SUMMARY:
RATIONALE: Diagnostic procedures, such as MRI and magnetic resonance spectroscopy imaging, may help in learning how well dutasteride works in patients with benign prostatic hypertrophy and low-risk prostate cancer.

PURPOSE: This clinical trial is studying MRI and magnetic resonance spectroscopy imaging in patients receiving dutasteride for benign prostatic hypertrophy and low-risk prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether there is a decrease in the extent of prostate cancer as measured by endorectal MRI and magnetic resonance spectroscopy imaging in patients with symptomatic benign prostatic hypertrophy and low-risk prostate cancer treated with dutasteride for 6 months.

Secondary

* To monitor the effects of dutasteride on serum testosterone, dihydrotestosterone, and free and total prostate-specific antigen (PSA).
* To monitor the effects of dutasteride on symptom and quality-of-life indices.

OUTLINE: Patients receive oral dutasteride once daily for 6 months.

Patients undergo endorectal MRI and magnetic resonance spectroscopy imaging at baseline and at 1, 3, and 6 months.

Patients complete quality-of-life questionnaires using the International Index of Erectile Function Questionnaire, American Urological Association Symptom Index, Functional Alterations due to Changes in Elimination, and Spitzer Quality-of-Life Index at baseline and at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed adenocarcinoma of the prostate

  * Clinical stage T1b, T1c, or T2a disease
  * Gleason score ≤ 6
  * Maximal prostate-specific antigen (PSA) < 10 ng/mL
* Demonstrates intra-prostatic metabolite abnormalities, consistent with adenocarcinoma of the prostate (i.e., ≥ 3 voxels with magnetic resonance spectroscopy imaging [MRSI] scores 4-5) by baseline MRI and MRSI
* Has symptomatic benign prostatic hypertrophy and is currently undergoing watchful waiting OR opting to undergo permanent seed implant (i.e., brachytherapy), but requires neoadjuvant androgen suppression for prostate shrinkage
* No regional lymph node involvement
* No evidence of distant metastases
* Zubrod performance status 0-1
* Able to swallow and retain oral medications

Exclusion Criteria:

* Other prior or concurrent invasive cancer, other than localized basal cell or squamous cell carcinoma of the skin
* Contraindications to MRI/MRSI, including any of the following:

  * Prostate biopsy (within the past 8 weeks) and any continued post-biopsy bleeding
  * Rectal bleeding
  * Anal fissures
  * Rectal surgery (end-to-end anastomosis)
  * Inflammatory bowel disease
  * Prior radical prostatectomy
  * Hip replacement
  * Certain types of penile implants
  * Vascular clips
  * Known anaphylactic reaction to latex compounds
  * Anticoagulant drugs
  * Severe claustrophobia
  * Cardiac pacemaker
  * Metal in eye
  * Any other metallic or foreign object in the body
* Unstable serious co-morbidities including, but not limited to, myocardial infarction, coronary artery syndrome, cardiac arrhythmias, symptomatic congestive heart failure, or cerebrovascular accident
* Major medical or psychiatric illness that, in the investigator's opinion, would preclude the completion of treatment and interfere with follow up
* Known hypersensitivity to any 5α-reductase inhibitor or drug chemically related to the study drug
* Prior radical surgery (prostatectomy) or cryosurgery for prostate cancer
* Prior pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* Prior or concurrent cytotoxic chemotherapy for prostate cancer
* Prior hormonal therapy, such as luteinizing hormone-releasing hormone agonists (e.g., goserelin or leuprolide acetate), antiandrogens (e.g., flutamide or bicalutamide), or estrogens (e.g., diethylstilbestrol)
* Prior or concurrent finasteride, dutasteride, other drugs with known antiandrogenic properties (e.g., spironolactone or progestational agents), or any dietary or herbal supplement (e.g., selenium, vitamin E, saw palmetto, or PC-SPES)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-06; Primary Completion 2008-12 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mack Roach, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from June 2005 to June 2008 from untreated patients seen at the University of California San Francisco
Groups:
- Dutasteride: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months
  dutasteride : 6 months of dutasteride 3.5 mg daily
Period: Overall Study
Arm/Group | Dutasteride
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dutasteride
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 65 [57 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10
Clinical Stage [Number; unit: Participants] — In the TNM system, T refers to the primary prostate tumor, N refers to the status of the lymph nodes near to the prostate, and M refers to the degree to which prostate cancer has traveled out of the immediate area of the prostate to other organs of the body (metastases). T1c = a positive prostate specific antigen (PSA) test but no other clinical sign of the disease (i.e., no abnormality felt on digital rectal examination or visible on any form of imaging test). T2a = tumor is palpable or visible on imaging (ultrasound or MRI) in not more than half of one side (one lobe) of the prostate.
  Participants
    T1c | 7
    T2a | 3
Total PSA [Median (Full Range); unit: ng/mL] — The prostate-specific antigen (PSA) test measures the blood level of PSA, a protein that is produced by the prostate gland.
  ng/mL | 5.05 [2.14 to 11.74]
Prostate volume [Mean (Full Range); unit: mL] — To assess prostate volume, regions of interest were manually drawn around the prostate across its full three-dimensional extent on the T2-weighted MR images; at subsequent timepoints, prostate volume was assessed as a percentage of the baseline value.
  mL | 47.3 [22.0 to 75.2]

OUTCOME MEASURES:

1. Primary Outcome: Change in Extent of Cancer
Description: Proportion of voxels consistent with prostate cancer as measured by magnetic resonance spectroscopy imaging (MRSI). MRSI spectra were examined and scored as healthy or cancerous. The change in cancerous volumes over time was evaluated. Because a significant decrease in citrate and polyamines on MRSI spectra was noted at 1 month compared with baseline, healthy tissue appeared to be more like cancer and thus created a false impression that the cancer had grown after 1 month. To reduce this bias, primary comparisons were made between the 1-month and 6-month scans.
Time Frame: 1 month, 6 months
Population: One participant withdrew from the study
Measure: Number; unit: participants
Arm/Group | Dutasteride
Number analyzed (Participants) | 9
participants
  30-45% Decrease | 3
  No change (95 - 100%) | 2
  65-167% Increase | 4

2. Secondary Outcome: Adverse Events Indicative of Safety of Dutasteride
Description: Toxicities from Dutasteride were recorded at each study visit and assessed by NCI-CTCAE v3.0.
Time Frame: Baseline, 1, 3, and 6 months
Measure: Number; unit: adverse events
Arm/Group | Dutasteride
Number analyzed (Participants) | 10
adverse events | 5

3. Secondary Outcome: Symptom Indices Over Time - IPSS
Description: IPSS (The International Prostate Symptom Score) is a symptom index based on seven questions concerning urinary symptoms (1 Incomplete emptying, 2 Frequency, 3 Intermittency, 4 Urgency, 5 Weak Stream, 6 Straining, 7 Nocturia) for which the patient chooses one out of six answers indicating increasing severity of the particular symptom, ranging from 0 (Not at all) to 5(Almost always). The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). Mild (symptom score less than of equal to 7); Moderate (symptom score range 8-19); Severe (symptom score range 20-35).
Time Frame: Baseline, 1, 3, and 6 months
Population: Because one participant withdrew from the study prior to 6-months, n=9 at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Dutasteride - Baseline: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. IPSS was assessed at Baseline.
- Dutasteride - 1 Month: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. IPSS was assessed at 1 month.
- Dutasteride - 3 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. IPSS was assessed at 3 months.
- Dutasteride - 6 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. IPSS was assessed at 6 months.
Arm/Group | Dutasteride - Baseline | Dutasteride - 1 Month | Dutasteride - 3 Months | Dutasteride - 6 Months
Number analyzed (Participants) | 10 | 10 | 10 | 9
units on a scale | 8.8 (3.8) | 6.6 (3.0) | 7.9 (4.4) | 5.9 (4.3)

4. Secondary Outcome: Symptom Indices Over Time - IIEF-5
Description: The International Index of Erectile Function (IIEF-5) is an abridged five-item version of the original IIEF 15-item questionnaire designed to evaluate erectile function, based on a definition arrived at by the National Institutes of Health Consensus Panel. Each of 5 questions about erectile function over the past 6 months is scored by the patient from 1 (severe dysfunction) to 5 (little or no dysfunction). The IIEF-5 is scored from 5 to 25, with lower scores indicating erectile dysfunction: 22-25 = No erectile dysfunction; 17-21 = Mild erectile dysfunction; 12-16 = Mild to moderate erectile dysfunction; 8-11 = Moderate erectile dysfunction; 5-7 = Severe erectile dysfunction
Time Frame: Baseline, 1, 3, and 6 months
Population: One participant withdrew from the study prior to the 6 month timepoint; thus n=9 at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Dutasteride - Baseline: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. IIEF-5 was assessed at baseline.
- Dutasteride - 1 Month: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. IIEF-5 was assessed at 1 month.
- Dutasteride - 3 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. IIEF-5 was assessed at 3 months.
- Dutasteride - 6 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. IIEF-5 was assessed at 6 months.
Arm/Group | Dutasteride - Baseline | Dutasteride - 1 Month | Dutasteride - 3 Months | Dutasteride - 6 Months
Number analyzed (Participants) | 10 | 10 | 10 | 9
units on a scale | 16.4 (7.8) | 17.0 (8.7) | 16.0 (7.9) | 15.3 (8.6)

5. Secondary Outcome: Health-Related Quality of Life (HRQL) Indices Over Time - FACE
Description: Functional Alterations due to Changes in Elimination (FACE) is a 14-item questionnaire designed to evaluate the effects of changes in urinary and bowel elimination on daily functioning. It is scored out of 56, with higher scores reflecting poorer HRQL.
Time Frame: Baseline, 1, 3, and 6 months
Population: One participant withdrew from the study prior to the 6 month timepoint; thus n=9 at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Dutasteride - Baseline: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. FACE was assessed at Baseline.
- Dutasteride - 1 Month: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. FACE was assessed at 1 month.
- Dutasteride - 3 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. FACE was assessed at 3 months.
- Dutasteride - 6 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. FACE was assessed at 6 months.
Arm/Group | Dutasteride - Baseline | Dutasteride - 1 Month | Dutasteride - 3 Months | Dutasteride - 6 Months
Number analyzed (Participants) | 10 | 10 | 10 | 9
units on a scale | 4.6 (2.5) | 4.7 (1.2) | 5.0 (1.9) | 4.8 (1.3)

6. Secondary Outcome: Health-Related Quality of Life (HRQL) Indices Over Time - SQLI
Description: The Spitzer Quality of Life Index (SQLI) is a validated five-item questionnaire evaluating global HRQL. Activity, daily living, health, support of family and friends, and outlook are each rated on a 3-point scale (0 to 2), with total score ranging from 0-10, with lower score indicating poorer HRQL.
Time Frame: Baseline, 1, 3, and 6 months
Population: One participant withdrew from the study prior to 6 months; thus, n=9 at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Dutasteride - Baseline: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. SQLI was assessed at Baseline.
- Dutasteride - 1 Month: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. SQLI was assessed at 1 month.
- Dutasteride - 3 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. SQLI was assessed at 3 months.
- Dutasteride - 6 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. SQLI was assessed at 6 months.
Arm/Group | Dutasteride - Baseline | Dutasteride - 1 Month | Dutasteride - 3 Months | Dutasteride - 6 Months
Number analyzed (Participants) | 10 | 10 | 10 | 9
units on a scale | 9.7 (0.7) | 9.9 (0.3) | 9.6 (0.7) | 9.9 (0.3)

7. Secondary Outcome: Total PSA Over Time
Time Frame: Baseline, 1, 3, and 6 months
Population: Because one participant withdrew from the study prior to 6-months, n=9 for the 6-month Mean(SD) levels.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dutasteride - Baseline: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. PSA was measured at Baseline.
- Dutasteride - 1 Month: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. PSA was measured at 1 month.
- Dutasteride - 3 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. PSA was measured at 3 months.
- Dutasteride - 6 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. PSA was measured at 6 months.
Arm/Group | Dutasteride - Baseline | Dutasteride - 1 Month | Dutasteride - 3 Months | Dutasteride - 6 Months
Number analyzed (Participants) | 10 | 10 | 10 | 9
ng/mL | 5.44 (2.90) | 4.33 (2.23) | 2.85 (1.49) | 2.59 (1.06)

8. Secondary Outcome: Dihydrotestosterone (DHT) Over Time
Time Frame: Baseline, 1, 3, and 6 months
Population: Because one participant withdrew from the study prior to 6-months, n=9 at 6 months.
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- Dutasteride - Baseline: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. DHT was measured at Baseline.
- Dutasteride - 1 Month: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. DHT was measured at 1 month.
- Dutasteride - 3 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. DHT was measured at 3 months.
- Dutasteride - 6 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. DHT was measured at 6 months.
Arm/Group | Dutasteride - Baseline | Dutasteride - 1 Month | Dutasteride - 3 Months | Dutasteride - 6 Months
Number analyzed (Participants) | 10 | 10 | 10 | 9
ng/dL | 33.5 (8.9) | 5.2 (5.5) | 2.5 (0.8) | 2.5 (0.8)

9. Secondary Outcome: Testosterone Over Time
Time Frame: Baseline, 1, 3, and 6 months
Population: Because one participant withdrew from the study prior to 6-months, n=9 at 6 months.
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- Dutasteride - Baseline: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. Testosterone was measured at Baseline.
- Dutasteride - 1 Month: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. Testosterone was measured at 1 month.
- Dutasteride - 3 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. Testosterone was measured at 3 months.
- Dutasteride - 6 Months: Dutasteride was administered at a dose of 3.5 mg as an oral soft gelatin capsule once daily for 6 months. Testosterone was measured at 6 months.
Arm/Group | Dutasteride - Baseline | Dutasteride - 1 Month | Dutasteride - 3 Months | Dutasteride - 6 Months
Number analyzed (Participants) | 10 | 10 | 10 | 9
ng/dL | 356.5 (109.3) | 418.4 (155.7) | 443.2 (132.1) | 484.3 (106.0)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Toxicities from dutasteride were recorded at each follow-up visit using the National Cancer Institute's Common Terminology Criteria for Adverse Events toxicity scale version 3.0
Arm/Group | Dutasteride
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dutasteride (N=10)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Decreased ejaculate volume (Reproductive system and breast disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The inclusion of only men with low volume disease may have limited our ability to accurately assess response rates after dutasteride due to the background effects on normal prostate metabolism.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes